CLINICAL TRIAL: NCT00933517
Title: Phase II Trial Assessing Neoadjuvant Therapy With FEC 100 Followed by Taxotere® (Docetaxel) Plus Vectibix® (Panitumumab) in Patients With Operable, HR and Her-2 Negative Breast Cancer. TVA Study
Brief Title: Assessment of the Efficacy of the Neoadjuvant Combination: "Chemotherapy-Targeted Therapy" in Breast Cancer.
Acronym: TVA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Getna7/CJP1.0
Record Dates: First submitted 2009-07-03; First posted 2009-07-07 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Pathological Response Rate
Keywords: breast cancer, neoadjuvant therapies, chemotherapy, targeted therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Panitumumab; Fluorouracil; Epirubicin; Cyclophosphamide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: vectibix — 9mg/kg at D1 of each 21-days cycle
Drug: fluorouracile — 500 mg/m2 at D1 of each 21-days cycle
Drug: Epirubicine — 100 mg/m2 at D1 of each 21-days cycle
Drug: cyclophosphamide — 500 mg/m2 at D1 of each 21 dyas cycle
Drug: docetaxel — 100 mg/m2 at D1 of each 21 days cycle

SUMMARY:
The purpose of this study is to assess the pathological response rate in operable breast cancer patients treated by neoadjuvant combination: "FEC-Taxotere/Vectibix".

ELIGIBILITY:
Inclusion Criteria:

* Age ³ 18.- Performance status £ 2 (according to WHO criteria).
* Patient has histologically confirmed, non-metastatic breast cancer, with a clinical tumour diameter of ³ 2 cm
* HR negative and Her-2 negative.
* Clinical stage II and IIIa.
* Patients not previously treated by surgery, radiotherapy, hormone therapy or chemotherapy.· Haematology: o Neutrophil count ≥1.5x109/Lo Platelet count ≥100x109/Lo Leucocyte count > 3,000/mmo Hb> 9g/dl· Hepatic Function:o Total bilirubin ≤ 1.5 time the upper normal limit (UNL)o ASAT ≤ 2.5xUNL in absence of liver metastases, or ≤5xUNL in presence of liver metastases ALAT ≤ 2.5xUNL in absence of liver metastases, or ≤5xUNL in presence of liver metastases Alkaline phosphatase ≤ 2.5 time the upper normal limit (UNL)· Renal Function· Creatinine clearance ≥50 mL/min and serum creatinine ≤1.5xUNL· Metabolic Function o Magnesium ≥ lower limit of normal. o Calcium ≥ lower limit of normal.
* Patient with no progressive heart disease, and for whom anthracyclines are not contraindicated (normal FEV).
* Patient has signed the consent forms for participation before inclusion in the trial.
* Member of a Social Security scheme (or a beneficiary of such a scheme) according to the provisions of the law of 9 August 2004.

Exclusion Criteria:

* Male patients.
* Her-2 positive patients
* Subject pregnant or breast feeding, or planning to become pregnant within 6 months after the end of treatment.
* Subject (male or female) is not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months (male or female) after the end of treatment.
* Any form of breast cancer other than those described in the inclusion criteria, particularly inflammatory and/or overlooked forms (T4b or T4d).
* Non-measurable tumour.
* Patients have already undergone surgery for their disease or have had primary axillary dissection.
* Patient has already been treated for new breast cancer.
* Patient is a ward.
* Patient has a history of second cancer, with exception of in situ cervical cancer or basocellular skin cancer which is regarded as cured.
* Patient has another disease which is deemed incompatible with the patient being included in the protocol.
* Heart or kidney failure, medullary, respiratory or liver failure.
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) £ 1 year before enrollment/randomization
* History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan
* Significant neurological or psychiatric abnormalities.
* Symptomatic or progressive disorder of the central nervous system (CNS) or metastasis at the initial check-up.
* Peripheral neuropathy > grade 2 (NCI-CTCAE criteria, Version 3.0).
* History of allergy to polysorbate 80.
* Concomitant treatment with a trial drug, participation in another clinical trial within < 30 days or previous chemotherapy.
* Patient with no fixed address in the next 6 months or living at a distance from the treatment centre so it is difficult to check her progress.
* Prior anti-EGFr antibody therapy (e.g.:cetuximab) or treatment with small molecule EGFr tyrosine kinase inhibitors (e.g.: erlotinib).
* Known previous or ongoing abuse of narcotic drug, other medication or alcohol.
* Any investigational agent within 30 days before initiation of study treatment. - Must not have had a major surgical procedure within 28 days of initiation of treatment.
* Subject unwilling or unable to comply with study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To assess the rate of complete histological response, according to Chevallier's classification | after 24 weeks of treatment

SECONDARY OUTCOMES:
the rate of complete histological response, according to Sataloff's classification; the rate of clinical, ultrasound, mammogram response, according to the WHO criteria; progression-free and overall survival; the tolerance. | After 24 weeks of treatment, at surgery and at five years

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - Centre Jean Perrin, Clermont-Ferrand, Clermont-Ferrand
  - Centre Paul Strauss, Strasbourg, Strasbourg
  - Pole Santé République, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - CHU Dupuytren, Limoges
  - Centre Léon Bérard, Lyon
  - Centre Hospitalier, Montluçon
  - Hôpital Tenon, Paris
  - Institut Jean Godinot, Reims
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Nabholtz JM, Abrial C, Mouret-Reynier MA, Dauplat MM, Weber B, Gligorov J, Forest AM, Tredan O, Vanlemmens L, Petit T, Guiu S, Van Praagh I, Jouannaud C, Dubray-Longeras P, Tubiana-Mathieu N, Benmammar KE, Kullab S, Bahadoor MR, Radosevic-Robin N, Kwiatkowski F, Desrichard A, Cayre A, Uhrhammer N, Chalabi N, Chollet P, Penault-Llorca F. Multicentric neoadjuvant phase II study of panitumumab combined with an anthracycline/taxane-based chemotherapy in operable triple-negative breast cancer: identification of biologically defined signatures predicting treatment impact. Ann Oncol. 2014 Aug;25(8):1570-7. doi: 10.1093/annonc/mdu183. Epub 2014 May 14. PMID 24827135